CLINICAL TRIAL: NCT05489120
Title: Randomized Controlled Trial of a Low-Protein Diet (LPD) With Low-Protein (LP) Foods Versus a LPD Without LP Foods in Patients With Chronic Kidney Disease (CKD): Efficacy and Feasibility Study
Brief Title: Low-Protein Diet With Low-Protein Foods Versus a LPD Without LP Foods in Patients With Chronic Kidney Disease (CKD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EFFLAVIS
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease Stage 3B; Chronic Kidney Disease stage4; Chronic Kidney Disease Stage 5; Chronic Kidney Disease Stage 3A
Keywords: low-protein diet; low-protein foods; FLAVIS; compliance; effectiveness; safety
MeSH Terms: conditions — Renal Insufficiency, Chronic; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COMPARATOR (No Intervention): Follow-up of the CKD patient according to current practice i.e. low protein diet.
- FLAVIS (Experimental): Follow-up of the CKD patient according to the current practice i.e. low protein diet with the addition of of low-protein products (FLAVIS).
  Interventions: Other: Consumption of FLAVIS

INTERVENTIONS:
Other: Consumption of FLAVIS — Patients of the FLAVIS group will recevied FLAVIS products in addition to their diet follow-up.
  Arms: FLAVIS

SUMMARY:
The KDOQI 2020 - Clinical practice guideline for nutrition in chronic kidney disease (CKD) -recommends protein restriction to reduce the risk of end-stage renal disease/death and improve quality of life, a low protein diet providing 0.55-0.60g dietary protein/ kg body weight/day is recommended. FLAVIS® is a product line of hypoprotein foods specially developed for the treatment of CKD.The use of low-protein foods may facilitate the achievement of nutritional goals in terms of protein intake and help patients to follow a low-protein diet.

ELIGIBILITY:
Inclusion Criteria:

* CKD patient stage 3a-5 (<60 ml/min/1.73 m² estimated by CKD-EPI formula) and not on dialysis,
* With a good nutritional status (i.e., absence of malnutrition according to albumin, pre-albumine, BMI and no clinical and paraclinical criteria of malnutrition),
* Above 1g protein/ kg bw (ideal body weight),
* LPD-naïve patient,
* Motivated to LPD introduction (ensure during screening phase patient willingness to modify diet habits with counselling accurate follow-up),
* Available to attend the visits planned by the protocol and able to complete the data collection documents (diet record and self-administered questionnaires),
* Subject affiliated to a health insurance system or is a beneficiary (art. L.1121-11, Code of Public Health, France),
* Having given their informed written consent regarding its participation to the protocol.

Exclusion Criteria:

* Patient for whom dialysis or transplantation is planned/expected within the next 12 months
* Known allergic reactions to the ingredients present in FLAVIS products (milk, eggs, soy, nut),
* Uncontrolled Diabetes (HbA1C >8.5%),
* Active cancer (including a 5 years remission period),
* Psychiatric disorders or inability to follow the protocol,
* Evidence of any active infectious or uncontrolled inflammatory diseases,
* Inability to provide blood samples (poor venous capital),
* Inability to perform correct 24-hours urine collection,
* Any change of the chronic medication within 1 month before screening,
* Presence of any significant medical finding or significant history such as uncontrolled systemic diseases that may impact the safety, the interpretation of the results and/or the participation of the subject in the study according to the opinion of the investigator,
* Patient with an active implanted medical device
* Simultaneous participation in another clinical trial or subject still within the exclusion period of a previous clinical trial.
* Vulnerable subjects (art. L. 1121-5 à 8 et L. 1122-1-2, Code of Public Health, France) are also excluded from the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2022-11-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Effectiveness in terms of protein intake of a LPD with LP foods (FLAVIS products) compared to standard products (LPD without consumption of LP foods) | 12 month
  Maroni formula : (Measurement of urea in urine + ([patient weight]*0.031))*6.25

SECONDARY OUTCOMES:
Protein intake during the 12 months follow-up | 1 month, 3 month, 6 month and 9 month
  Maroni formula: (Measurement of urea in urine + ([patient weight]*0.031))*6.25
Dietary adherence | baseline, 1 month, 3 month, 6 month and 12 month
  3-day dietary record correlated to a 24-hour urine collection
Dietary compliance for products under study | monthly up to 12 months
  quantities consumed of FLAVIS products.
Effects of the LPD on BMI | baseline, 1 month, 3 month, 6 month and 12 month
  Weight and height will be combined to report BMI in kg/m^2.
Effects of the LPD on weight | baseline, 1 month, 3 month, 6 month and 12 month
  Weight in kg
Effects of the LPD on body composition: water | baseline, 1 month, 3 month, 6 month and 12 month
  Water in litres
Effects of the LPD on body composition: muscles | baseline, 1 month, 3 month, 6 month and 12 month
  Muscles in Kg
Effects of the LPD on body composition: body protein content | baseline, 1 month, 3 month, 6 month and 12 month
  Body protein content in Kg
Effects of the LPD on Blood | baseline, 1 month, 3 month, 6 month, 9 month and 12 month
  Blood Chemistry
Effects of the LPD on Urine | baseline, 1 month, 3 month, 6 month, 9 month and 12 month
  Urine Chemistry
Effects of the LPD on diabetic patient glycemic profile | Baseline, 6 month and 12 month
  Hb1Ac will be measured
Incidence of Adverse Events [Safety of the LPD] | 1 month, 3 month, 6 month, 9 month and 12 month
  Questioning and a clinical examination, biological analyses review
Incidence of Adverse Events [Safety of the LPD] | 3 month, 6 month and 12 month
  4-points Likert scale
Patient quality of life | baseline, 3 month, 6 month and 12 month
  SF-36 questionnaire score which from 0 to 100
Patient satisfaction with LPD | 3 month, 6 month and 12 month
  Auto-questionnaire with numerical scales, closed-ended questions and Likert scales

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Koppe, Dr, Study Director — HCL
Locations (21):
- France (21):
  - Clinique sainte isabelle, Abbeville
  - Cabinet médical du Dr Magnant, Aix-en-Provence
  - CHU Besançon, Besançon
  - Maison du Rein, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH Chalon, Chalon-sur-Saône
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Santélys BFC, Dijon
  - CH Le Mans, Le Mans
  - Hospices Civiles de Lyon, Lyon
  - Hôpital Edouard Heriot, Lyon
  - Saint Joseph Saint Luc, Lyon
  - Hôpital la conception, Marseille
  - CH Mâcon, Mâcon
  - APHP - Hôpital Necker, Paris
  - AURA Paris, Paris
  - Tenon hospital -APHP, Paris
  - Hôpital Drôme Nord, Romans-sur-Isère
  - Nouvel Hôpital Civil, Strasbourg
  - Calydial, Vienne
  - Hôpital Nord-Ouest, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No